CLINICAL TRIAL: NCT01743027
Title: Phase 3, Efficacy and Safety Study of AL-4943A Ophthalmic Solution, 0.77% in Patients With Allergic Conjunctivitis Using the Conjunctival Allergen Challenge (CAC) Model
Brief Title: Efficacy and Safety of an Ophthalmic Solution in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-053
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis; Olopatadine HCl solution; Conjunctival Allergen Challenge; Itching eyes; Ocular allergies; PATADAY; PATANOL
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AL-4943A (Experimental): AL-4943A ophthalmic solution, 1 drop per eye Day 0, followed by 1 drop per eye Day 14
  Interventions: Drug: AL-4943A ophthalmic solution
- PATADAY (Active Comparator): Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop per eye Day 0, followed by 1 drop per eye Day 14
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%
- PATANOL (Active Comparator): Olopatadine hydrochloride ophthalmic solution, 0.1%, 1 drop per eye Day 0, followed by 1 drop per eye Day 14
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.1%
- Vehicle (Placebo Comparator): AL-4943A ophthalmic solution vehicle, 1 drop per eye Day 0, followed by 1 drop per eye Day 14
  Interventions: Drug: AL-4943A ophthalmic solution vehicle

INTERVENTIONS:
Drug: AL-4943A ophthalmic solution
  Arms: AL-4943A
Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%
  Other Names: PATADAY®
  Arms: PATADAY
Drug: Olopatadine hydrochloride ophthalmic solution, 0.1%
  Other Names: PATANOL®
  Arms: PATANOL
Drug: AL-4943A ophthalmic solution vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate an ophthalmic solution for the treatment of ocular itching associated with allergic conjunctivitis using the Conjunctival Allergen Challenge (CAC) model.

DETAILED DESCRIPTION:
Enrolled participants will be tested for the presence of common allergies using the Conjunctival Allergen Challenge (CAC) model. Drops of increasing concentration of a solubilized allergen will be instilled in both eyes until a positive reaction occurred. The test will be repeated to confirm the allergic reaction. Participants with confirmed reactions will be administered the test article (Day 0) and undergo a CAC 24 hours post-instillation (Day 1). On Day 14, participants will be administered the test article and undergo an additional CAC.

ELIGIBILITY:
Inclusion Criteria:

* Able to be dosed in both eyes, able and willing to make the required study visits and to follow instructions.
* Negative urine pregnancy test if female of childbearing potential and use adequate birth control throughout the study period.
* Diagnostic skin test indicative of allergy for cat hair, cat dander, grasses, ragweed, dust mite, dog dander, cockroach and/or trees within 24 months prior to Visit 1 or at Visit 1.
* History of seasonal or perennial allergic conjunctivitis for at least 1 year prior to Visit 1.
* Best-corrected visual acuity of 55 or greater in each eye as measured by ETDRS (letters read method).
* Manifest a positive bilateral Conjunctival Allergen Challenge (CAC) test response.
* Willing to discontinue contact lens wear for at least 72 hours prior to Visit 1 and throughout the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known history or presence of persistent dry eye syndrome, or currently requires frequent use of artificial tears, gels or lubricants, presence of punctal plugs, use of Restasis®, or topical ocular corticosteroids for dryness of eyes.
* Presence of an ocular condition that may affect the study outcomes.
* History or evidence of ocular surgery (including refractive procedures such as LASIK, PRK and RK) within 6 months of Visit 1.
* Presence of signs/symptoms of active allergic conjunctivitis at the start of Visits 1, 2, 3A, or 4.
* History of anaphylactic reaction to any allergens used in this study.
* Current evidence or recent (within 6 months) history of severe, unstable, or uncontrolled medical conditions and/or other relevant systemic diseases.
* Use of any disallowed medication without protocol-specified washout period prior to Visit 1, or during the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Narvekar, MS, MBBS, Study Director — Alcon Research

REFERENCES:
- [Derived] Carr W, Schaeffer J, Donnenfeld E. Treating allergic conjunctivitis: A once-daily medication that provides 24-hour symptom relief. Allergy Rhinol (Providence). 2016 Jan;7(2):107-14. doi: 10.2500/ar.2016.7.0158. Epub 2016 Jul 26. PMID 27466061
- [Derived] McLaurin E, Narvekar A, Gomes P, Adewale A, Torkildsen G. Phase 3 Randomized Double-Masked Study of Efficacy and Safety of Once-Daily 0.77% Olopatadine Hydrochloride Ophthalmic Solution in Subjects With Allergic Conjunctivitis Using the Conjunctival Allergen Challenge Model. Cornea. 2015 Oct;34(10):1245-51. doi: 10.1097/ICO.0000000000000562. PMID 26266427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 study centers located in the US.
Pre-assignment Details: Of the 902 enrolled, 557 participants discontinued prior to randomization due to screen failure (390), adverse event (12), lost to follow-up (26), protocol violation (2), withdrawal by patient (85), and other (42). This reporting group includes all randomized participants (345).
Period: Overall Study
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Started | 98 | 99 | 99 | 49
Completed | 93 | 94 | 90 | 48
Not Completed | 5 | 5 | 9 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 1 | 4 | 3 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle | Total
Number analyzed (Participants) | 98 | 99 | 99 | 49 | 345
Age, Customized [Number; unit: participants]
  18-64 Years | 97 | 93 | 95 | 48 | 333
  ≥65 - <75 Years | 1 | 5 | 4 | 1 | 11
  ≥75 - <85 Years | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 55 | 56 | 32 | 204
  Male | 37 | 44 | 43 | 17 | 141

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Itching at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop installation. Ocular itching was assessed by the participant on a 0-4 scale (0= none, 4 = incapacitating itch). Average of ocular itching score over both eyes was analyzed.
Time Frame: Day 14 (3, 5, and 7 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  3 minutes post-CAC | 0.38 (0.069) | 0.47 (0.069) | 0.59 (0.070) | 1.91 (0.095)
  5 minutes post-CAC | 0.53 (0.075) | 0.61 (0.075) | 0.79 (0.076) | 1.99 (0.103)
  7 minutes post-CAC | 0.65 (0.081) | 0.61 (0.082) | 0.83 (0.083) | 1.82 (0.113)

2. Primary Outcome: Mean Ocular Itching at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation on Day 0. Ocular itching was assessed by the participant on a 0-4 scale (0= none, 4 = incapacitating itch). Average of ocular itching score over both eyes was analyzed.
Time Frame: Day 1 (3, 5, and 7 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  3 minutes post-CAC | 1.01 (0.093) | 1.33 (0.093) | 1.53 (0.093) | 2.30 (0.132)
  5 minutes post-CAC | 1.22 (0.092) | 1.48 (0.092) | 1.70 (0.091) | 2.37 (0.130)
  7 minutes post-CAC | 1.25 (0.097) | 1.41 (0.097) | 1.64 (0.096) | 2.14 (0.137)

3. Secondary Outcome: Mean Conjunctival Redness at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop installation. Conjunctival redness was assessed by the investigator on a 0-4 scale (0=none, 4=extremely severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: Day 14 (7, 15, and 20 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  7 minutes post-CAC | 1.34 (0.082) | 1.62 (0.082) | 1.65 (0.083) | 1.96 (0.113)
  15 minutes post-CAC | 1.65 (0.082) | 1.96 (0.082) | 1.97 (0.083) | 2.10 (0.112)
  20 minutes post-CAC | 1.66 (0.082) | 1.97 (0.082) | 1.97 (0.083) | 2.15 (0.113)

4. Secondary Outcome: Mean Conjunctival Redness at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation on Day 0. Conjunctival redness was assessed by the investigator on a 0-4 scale (0=none, 4=extremely severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: Day 1 (7, 15, and 20 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  7 minutes post-CAC | 1.92 (0.074) | 2.01 (0.073) | 1.97 (0.073) | 2.09 (0.104)
  15 minutes post-CAC | 2.04 (0.073) | 2.21 (0.073) | 2.10 (0.073) | 2.22 (0.104)
  20 minutes post-CAC | 2.08 (0.078) | 2.19 (0.078) | 2.07 (0.077) | 2.23 (0.110)

5. Secondary Outcome: Mean Total Redness at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop installation. Conjunctival redness, ciliary redness, and episcleral redness were assessed by the investigator on 0-4 scale (0=none, 4=extremely severe). Total redness is a composite variable summing conjunctival redness, ciliary redness, and episcleral redness scores (resultant score 0-12). The average of total redness over both eyes was analyzed.
Time Frame: Day 14 (7, 15, and 20 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  7 minutes post-CAC | 3.92 (0.239) | 4.73 (0.240) | 4.82 (0.243) | 5.93 (0.330)
  15 minutes post-CAC | 4.80 (0.240) | 5.73 (0.240) | 5.85 (0.243) | 6.50 (0.330)
  20 minutes post-CAC | 4.96 (0.244) | 5.88 (0.245) | 5.88 (0.248) | 6.67 (0.337)

6. Secondary Outcome: Mean Total Redness at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation on Day 0. Conjunctival redness, ciliary redness, and episcleral redness were assessed by the investigator on 0-4 scale (0=none, 4=extremely severe). Total redness is a composite variable summing conjunctival redness, ciliary redness, and episcleral redness scores (resultant score 0-12). The average of total redness over both eyes was analyzed.
Time Frame: Day 1 (7, 15, and 20 minutes post-CAC)
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
units on a scale
  7 minutes post-CAC | 5.39 (0.214) | 5.77 (0.213) | 5.66 (0.212) | 6.12 (0.302)
  15 minutes post-CAC | 5.87 (0.216) | 6.42 (0.215) | 6.11 (0.215) | 6.49 (0.306)
  20 minutes post-CAC | 6.00 (0.230) | 6.41 (0.228) | 6.02 (0.228) | 6.49 (0.325)

7. Secondary Outcome: Proportion of Ocular Itching Responders at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop installation. Ocular itching was assessed by the participant on a 0-4 scale (0= none, 4 = incapacitating itch). A responder was defined as a participant with zero-itch (a score of zero on ocular itching for both eyes) or with at least 2 units reduction in ocular itching relative to the baseline confirmatory CAC score. Ocular itching score was averaged across both eyes and over the 3 post-CAC assessments (3, 5, and 7 minutes) for the calculation of units reduction. Proportion of Ocular Itching Responders is reported as a percentage.
Time Frame: Day 14
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication. Patients with missing data were considered as nonresponders in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
percentage of participants | 71.4 | 73.7 | 59.6 | 10.2

8. Secondary Outcome: Proportion of Itch Responders at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation on Day 0. Ocular itching was assessed by the participant on a 0-4 scale (0= none, 4 = incapacitating itch). A responder was defined as a participant with zero-itch (a score of zero on ocular itching for both eyes) or with at least 2 units reduction in ocular itching relative to the baseline confirmatory CAC score. Ocular itching score was averaged across both eyes and over the 3 post-CAC assessments (3, 5, and 7 minutes) for the calculation of units reduction. Proportion of Ocular Itching Responders is reported as a percentage.
Time Frame: Day 1
Population: Intent to Treat (ITT): This analysis population includes all randomized patients who received study medication.Patients with missing data were considered as nonresponders in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Number analyzed (Participants) | 98 | 99 | 99 | 49
percentage of participants | 40.8 | 30.3 | 26.3 | 4.1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (6 months). This analysis population includes all participants who were exposed to investigational product for 1-2 instillation(s).
Description: An adverse event was defined as any untoward medical occurrence in a patient who was administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Reports of AEs were obtained as solicited comments from the study patients and as observations by the study Investigator.
Arm/Group | AL-4943A | PATADAY | PATANOL | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/99 | 0/99 | 0/49
Other Adverse Events (participants affected / at risk) | 0/98 | 0/99 | 0/99 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.